CLINICAL TRIAL: NCT03757754
Title: Evalution of Safety, Tolerability and Pharmacokinetics of of HPPH in Ascending Dose for Cancer Patients in Phase I Clinical Trial
Brief Title: HPPH Photodynamic Therapy for Patients With Esophageal Cancer
Acronym: HPPH
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhejiang Hisun Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HISUN-HPPH-I-2014
Record Dates: First submitted 2018-10-22; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Esophageal Cancer
Keywords: PHHP; Esophageal cancer; Phase I study
MeSH Terms: conditions — Esophageal Neoplasms | interventions — 2-(1-hexyloxyethyl)-2-devinyl pyropheophorbide-a

STUDY DESIGN:
Intervention Model Description: Multiple Ascending Dose, Multiple groups, Multiple centers
Masking Description: open
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- HPPH 2.5 mg/m2 (Experimental): HPPH 2.5 mg/m2, Freeze-dried powder injection, intravenous infusion once daily, and a fixed light dose of 150 J/cm delivered 48 hours after infusion of HPPH.
  Interventions: Drug: HPPH 2.5 mg/m2
- HPPH 3 mg/m2 (Experimental): HPPH 3 mg/m2, Freeze-dried powder injection, intravenous infusion once daily, and a fixed light dose of 150 J/cm delivered 48 hours after infusion of HPPH.
  Interventions: Drug: HPPH 3 mg/m2
- HPPH 3.5 mg/m2 (Experimental): HPPH 3.5 mg/m2, Freeze-dried powder injection, intravenous infusion once daily, and a fixed light dose of 150 J/cm delivered 48 hours after infusion of HPPH.
  Interventions: Drug: HPPH 3.5 mg/m2
- HPPH 4 mg/m2 (Experimental): HPPH 4 mg/m2, Freeze-dried powder injection, intravenous infusion once daily, and a fixed light dose of 150 J/cm delivered 48 hours after infusion of HPPH.
  Interventions: Drug: HPPH 4 mg/m2
- HPPH 5 mg/m2 (Experimental): HPPH 5 mg/m2, Freeze-dried powder injection, intravenous infusion once daily, and a fixed light dose of 150 J/cm delivered 48 hours after infusion of HPPH.
  Interventions: Drug: HPPH 5 mg/m2
- HPPH 6 mg/m2 (Experimental): HPPH 6 mg/m2, Freeze-dried powder injection, intravenous infusion once daily, and a fixed light dose of 150 J/cm delivered 48 hours after infusion of HPPH.
  Interventions: Drug: HPPH 6 mg/m2

INTERVENTIONS:
Drug: HPPH 2.5 mg/m2 — HPPH was administered as a single, 2.5 mg/m2, slow intravenous infusion over 1 hour , and a fixed light dose of 150 J/cm delivered 48 hours after infusion of HPPH.
  Arms: HPPH 2.5 mg/m2
Drug: HPPH 3 mg/m2 — HPPH was administered as a single, 3 mg/m2, slow intravenous infusion over 1 hour, and a fixed light dose of 150 J/cm delivered 48 hours after infusion of HPPH.
  Arms: HPPH 3 mg/m2
Drug: HPPH 3.5 mg/m2 — HPPH was administered as a single, 3.5 mg/m2, slow intravenous infusion over 1 hour, and a fixed light dose of 150 J/cm delivered 48 hours after infusion of HPPH.
  Arms: HPPH 3.5 mg/m2
Drug: HPPH 4 mg/m2 — HPPH was administered as a single, 4 mg/m2, slow intravenous infusion over 1 hour, and a fixed light dose of 150 J/cm delivered 48 hours after infusion of HPPH.
  Arms: HPPH 4 mg/m2
Drug: HPPH 5 mg/m2 — HPPH was administered as a single, 5 mg/m2, slow intravenous infusion over 1 hour, and a fixed light dose of 150 J/cm delivered 48 hours after infusion of HPPH.
  Arms: HPPH 5 mg/m2
Drug: HPPH 6 mg/m2 — HPPH was administered as a single, 6 mg/m2, slow intravenous infusion over 1 hour, and a fixed light dose of 150 J/cm delivered 48 hours after infusion of HPPH.
  Arms: HPPH 6 mg/m2

SUMMARY:
Phase I study was to investigate the safety and tolerability of the photosensitizer (PS) 2-[1-hexyloxyethyl]-2-devinyl pyropheophorbide-a (HPPH) for injection in patients with Esophageal Cancer. It was to characterize the pharmacokinetics of HPPH and efficacy of HPPH.

DETAILED DESCRIPTION:
The present study is phase I study to evaluate the safety, tolerability, and pharmacokinetics of multiple ascending injection doses of HPPH in Patients with Esophageal Cancer. Up to 30 patients are planned to be enrolled in 6 cohorts with each cohort consisting of 3-6 patients ( male and/or female patients). In each cohort, patients will receive HPPH and Lyophilized treatment. The dose escalation in Cohorts was from 2.5 to 3, 3.5, 4, 5, and 6mg/m2 of HPPH, respectively, administered intravenous drop infusion over 1 hour, once daily, and a fixed light dose of 150 J/cm delivered 48 hours after infusion of HPPH.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, Male and female subjects with practicing a highly effective form of birth control, and a signed consent;
* Subjects who was diagnosed as Esophageal Cancer or carcinoma of gastric cardia by endoscopy and Biopsy pathology at T1-T3 stage.
* Subjects who could not be taken surgery or chemotherapy; with unsucessful surgery or failed chemotherapy; who had refused surgery and chemotherapy
* ECOG 0-2, Life expectancy would be more than 3-month

Exclusion Criteria:

* Subjects were diagnosed as Tracheoesophageal fistula or Esophageal mediatinal fistula, or more than 60 years old with having three kinds of Heart, Lung, Liver and Kidney commorbities;
* Hematopoietic WBC < 3×109/L; HGB <80g/L; PLT <80×109/L; PLT <1.5 times upper limit of normal (ULN)
* Hepatic TBIL>1.5ULN, ALT or AST >2.5 ULN
* Alkaline phosphatase > 3 times ULN
* Uncontrol Hypertension: Bp>160/100mmHg
* Uncomtrol Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-06-03 (Actual); Primary Completion 2019-01-20 (Estimated); Study Completion 2019-05-27 (Estimated)

PRIMARY OUTCOMES:
The number of dose-limiting toxicity | Day 1 to Day 10
  Dose-limiting toxicity would be assesed by CTCAE4.0

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | Day 1 to Day 84
  PK measurement expressed as Cmax for HPPH
Time to maximum concentration (tmax) | Day 1 to Day 84
  PK measurement expressed as Tmax for HPPH
Apparent terminal elimination phase half (t1/2) | Day 1 to Day 84
  PK measurement expressed as t1/2 for HPPH
Area under the concentration-time curve over the dosing interval (AUC0-t) | Day 1 to Day 84
  PK measurement expressed as AUC0-t for HPPH
Area under the concentration-time curve from zero extrapolated to infinity (AUC0-∞) | Day 1 to Day 84
  PK measurement expressed as AUC0-∞ for HPPH

CONTACTS AND LOCATIONS:
Overall Officials: Huilong Liu, PhD, Principal Investigator — General Hospital of Beijing Miitary Command of PLA
Locations (1):
- Department of Oncology, General Hospital of Beijing Miitary Command of PLA, Beijing, Beijing Municipality, China